CLINICAL TRIAL: NCT00030420
Title: Evaluation Of Celecoxib In Combination With Docetaxel In The Treatment Of Advanced Non-Small Cell Lung Cancer Patients Previously Treated With Platinum Based Chemotherapy
Brief Title: Celecoxib and Docetaxel in Treating Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069164; P30CA022453 (NIH); WSU-C-2304 (Other: Barbara Ann Karmanos Cancer Institute); NCI-V01-1688
Record Dates: First submitted 2002-02-14; First posted 2003-10-21 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Celecoxib & Docetaxel (Experimental): Celecoxib: 400mg by mouth, twice a day, each dose given with meals, to start -7 days prior to first cycle of treatment.
  Doctaxel: Day 1, 75mg/m2 IV over 60 minutes, repeated every 21 days
  Interventions: Drug: Celecoxib; Drug: Docetaxel

INTERVENTIONS:
Drug: Celecoxib — 400mg by mouth, twice a day, each dose given with meals, to start -7 days prior to first cycle of treatment.
  Other Names: Celebrex; Celebra; Onsenal
Drug: Docetaxel — On day 1, 75mg/m2 IV over 60 minutes, repeated every 21 days
  Other Names: Taxotere

SUMMARY:
RATIONALE: Celecoxib may slow the growth of cancer by stopping blood flow to the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with celecoxib may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining celecoxib and docetaxel in treating patients who have advanced non-small cell lung cancer that has been previously treated with platinum-based chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy and feasibility of celecoxib combined with docetaxel in patients with advanced non-small cell lung cancer previously treated with platinum-based chemotherapy.
* Determine the response rate of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral celecoxib twice daily (beginning on day -7 of the first course) and docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) receive 2 additional courses after CR. Patients who achieve stable disease (SD) or a partial response (PR) receive a minimum of 2 additional courses after SD or PR. At the discretion of the treating physician, patients then receive maintenance therapy comprising celecoxib only.

Patients who discontinue therapy for disease progression or unacceptable toxicity are followed for at least 6 months.

PROJECTED ACCRUAL: A total of 21-39 patients will be accrued for this study within 13-28 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage IIIA, IIIB, or IV non-small cell lung cancer

  * Disease progression during or after 1 or more platinum-based chemotherapy regimens
* Measurable or evaluable disease
* No symptomatic or untreated brain or leptomeningeal metastases

  * Previously treated patients must be neurologically stable for 4 weeks after completion of appropriate therapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* AST/ALT no greater than ULN (or no greater than 2.5 times ULN if alkaline phosphatase no greater than ULN)
* Alkaline phosphatase no greater than ULN (or no greater than 5 times ULN if AST/ALT no greater than ULN)
* No history of chronic hepatitis of any duration

Renal:

* Creatinine no greater than ULN

Cardiovascular:

* No uncontrolled congestive heart failure
* No uncontrolled angina
* No myocardial infarction and/or stroke within the past 6 months
* No active thromboembolic event within the past 4 weeks

Gastrointestinal:

* No gastrointestinal bleeding within the past 6 months
* No history of peptic ulcer disease

Other:

* No prior hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No prior allergy to any non-steroidal anti-inflammatory drug
* No other prior or concurrent malignancy within the past 3 years except adequately treated squamous cell or basal cell skin cancer or carcinoma in situ of the cervix
* No grade 2 or greater peripheral neuropathy
* No active infection
* No other serious concurrent medical illness
* No history of dementia, active psychiatric disorder, or other condition that would interfere with ability to take oral medication or preclude compliance with study
* HIV negative
* Must weigh at least 50 kg (110 pounds)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* Prior paclitaxel allowed
* No prior docetaxel

Endocrine therapy:

* At least 3 days since prior steroids

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to target lesion

Surgery:

* At least 4 weeks since prior major surgery

Other:

* Prior intermittent use of non-steroidal anti-inflammatory drugs (NSAIDs), including rofecoxib or celecoxib, allowed
* At least 1 week since prior fluconazole
* No recent prior NSAIDs, including rofecoxib or celecoxib, for a duration of more than 30 consecutive days
* No concurrent fluconazole or lithium
* No other concurrent NSAIDs except aspirin administered at a dose of no more than 325 mg/day for cardiovascular conditions
* No other concurrent cyclo-oxygenase-2 inhibitors
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2001-10; Primary Completion 2004-05 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of combining Celecoxib with Docetaxel | Weeks 1 , 2 and 3
  Blood levels of VEGF & PGE2

SECONDARY OUTCOMES:
Response rate of Celecoxib and Docetaxel | Every 2 cycles (or every 42 days); After therapy is completed or if the patient is only on Celecoxib, will be assessed for progression every month by clinical exam and every 3 months by radiological evaluation.
  CT Chest/Abdomen
Toxicity of Celecoxib and Docetaxel | Every week
  Routine bloodwork
Expression of cyclooxygenase-2 (COX-2) in tumors | Pre-study
  Tissue sample from initial diagnosis, parrafin embedded tissue block
Changes in plasma levels of prostaglandin E2 (PGE2) & vascular endthelial growth factor (VEGF) | Pre-study; Weeks 1 , 2 and 3
  Collecting blood plasma
Vascular changes induced in the tumor by celecoxib | Weeks 1, 3 & 6
  Using DCE-MRI and PET scans to evaluate.

CONTACTS AND LOCATIONS:
Overall Officials: Shirish M. Gadgeel, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Result] Schneider BJ, Kalemkerian GP, Kraut MJ, Wozniak AJ, Worden FP, Smith DW, Chen W, Gadgeel SM. Phase II study of celecoxib and docetaxel in non-small cell lung cancer (NSCLC) patients with progression after platinum-based therapy. J Thorac Oncol. 2008 Dec;3(12):1454-9. doi: 10.1097/JTO.0b013e31818de1d2. PMID 19057272